CLINICAL TRIAL: NCT06935864
Title: The Prognostic Value of Tissue Expression of Krüppel-Like Factors 4 and 7 in Bone Tumors
Brief Title: Tissue Expression of Krüppel-Like Factors 4 and 7 in Bone Tumors
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD173/2024; FMASU MD173/2024 (Other: Faculty of Medicine Ain Shams University Research Ethical Committee)
Record Dates: First submitted 2025-01-05; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Osteosarcoma in Children; Ewing Sarcoma of Bone or Soft Tissue
Keywords: Bone Tumor; Osteosarcoma; Ewing sarcoma
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective Arm: Children, young adolescents younger than 15 years, and young adults (15 to 39 years) with histologically confirmed patients with skeletal or extra-skeletal OS or ES with localized or metastatic disease stages.
  Interventions: Diagnostic Test: KLF factor (4 and 7)

INTERVENTIONS:
Diagnostic Test: KLF factor (4 and 7) — Immunohistochemical staining of 4 um sections prepared from paraffin blocks using KLF factor (4 and 7) by automated immunostaining using the streptavidin-biotin technique.

SUMMARY:
The current study is to assess the prognostic value of Krüppel-like factors 4 and 7 in bone tumors, and its role in the disease progression.

DETAILED DESCRIPTION:
Krüppel-like factors are a group of proteins that engage in different cell functions including proliferation, apoptosis, autophagy, invasion, and migration, and have been discovered to play an important role in bone disease development.

Study Setting: Pediatric Hematology, Oncology and Bone Marrow Transplantation Unit at Ain Shams University Children's Hospital.

* Type of Study: Prospective cohort.
* Study Period: 12 months.
* Study Population: Children, adolescents, and young adults diagnosed with localized and metastatic both skeletal and extra-skeletal osteosarcoma and Ewing's sarcoma
* Sampling Method: Convenience
* The medical history by direct interview of participants or from the patients files with a focus on:

  * Symptoms such as pain, swelling, and fracture including duration, intensity, and timing of complaint.
  * Specific events for bone tumors include prior benign/malignant lesions, family history, and previous radiotherapy for a prior cancer.
  * Assessment of the adverse outcomes.
  * Treatment protocol, timing of local control, type of local surgical control, need for adjuvant or definitive radiation therapy.
* Examination carried out upon initial patients' presentation (collected from files in the historical group):

  * A full physical examination including weight and height, with calculation of body mass index (BMI) and surface area (SA).
  * Local examination with specific attention to the size, consistency of the swelling, its location and mobility, the relation of swelling to the involved bone, and the presence of regional/ local lymph nodes.
* Radiologic investigations at initial diagnosis, after induction chemotherapy, after local control, as well as at the end of therapy and every 3 months during 1st 2 years after therapy (collected from files in the historical group):

  * Conventional radiographs in two planes
  * Magnetic resonance imaging (MRI) of the whole compartment with adjacent joints,
  * Computed tomography (CT) should be used only in the case of diagnostic problems or doubt, to visualize more clearly calcification, periosteal bone formation, or cortical destruction
  * Stage classification: positron emission tomography (PET)/CT using General Electric device number 5632.
* Laboratory assessment at presentation for cohort group (collected from files in the historical group)

  * Complete blood count (CBC)
  * Electrolytes including serum Calcium, phosphorus, magnesium, bicarbonate; creatinine, blood urea nitrogen, liver enzymes, and lactate dehydrogenase (LDH)
* Pathological methods:

  * Histopathological examination of H&E-stained sections prepared from paraffin blocks at 4-5 um thickness.
  * Immunohistochemical staining of 4 um sections prepared from paraffin blocks using KLF factor (4 and 7); this will be done with automated immunostaining using the streptavidin-biotin technique.
  * Interpretation of the stained slides will be done using a semiquantitative score and the results will be statistically analyzed.
* Sample Size: 30 patients

ELIGIBILITY:
Inclusion Criteria:

Age: children, young adolescents younger than 15 years, and young adults (15 to 39 years) Gender: Males and female. Histologically confirmed patients with skeletal or extra-skeletal OS or ES. Both localized and metastatic disease stages.

Exclusion Criteria:

Patients with second malignant bone sarcoma. Patients with benign bone tumors.

Ages: 1 Month to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults diagnosed with localized and metastatic both skeletal and extra-skeletal osteosarcoma and Ewing's sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The prognostic value | 1 year
  Assess the prognostic value of Krüppel-like factors 4 and 7 in bone tumors,

CONTACTS AND LOCATIONS:
Overall Officials: Fatma S E Ebeid, Principal Investigator — Faculty of Medicine Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo
  - Faculty of Medicine Ain Shams Research Institute- Clinical Research Center (MASRI-CRC), Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10977429/